CLINICAL TRIAL: NCT02531126
Title: A Phase 3, Multicenter, Open-Label Extension Trial of Oral RPC1063 as Therapy for Moderate to Severe Ulcerative Colitis
Brief Title: An Extension Study of RPC1063 as Therapy for Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPC01-3102; 2015-001600-64 (EudraCT Number); U1111-1218-0284 (Registry Identifier: WHO)
Record Dates: First submitted 2015-08-20; First posted 2015-08-24 (Estimated); Results first posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ozanimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RPC0163 (Ozanimod) (Experimental)
  Interventions: Drug: RPC1063

INTERVENTIONS:
Drug: RPC1063
  Other Names: Ozanimod

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of RPC1063 in participants with moderately to severely active ulcerative colitis. Only those participants who have previously participated in a trial of RPC1063, being either RPC01-3101 or completed at least 1 year of the open-label period of RPC01-202 will be eligible.

DETAILED DESCRIPTION:
This is an extension study trial. Eligible participants from the RPC01-3101 and RPC01-202 trials were able to roll-over in this trial to receive study medication until March 2023 or until the Sponsor discontinues the development program, whichever comes first.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit: www.BMSStudyConnect.com

Inclusion Criteria:

• Previously participated in a trial of RPC1063 and meets the criteria for participation in the open-label extension as outlined in the prior trial

Exclusion Criteria:

* Receiving treatment with breast cancer resistance protein inhibitors
* Clinically relevant cardiovascular conditions
* Liver function impairment

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 877 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (41):
- United States (10):
  - Local Institution - 144, Tucson, Arizona
  - Local Institution - 102, Anaheim, California
  - Local Institution - 117, Mission Hills, California
  - Local Institution - 112, Oak Lawn, Illinois
  - Local Institution - 119, Baton Rouge, Louisiana
  - Local Institution - 127, Jacksonville, North Carolina
  - Local Institution - 290, Oklahoma City, Oklahoma
  - Local Institution - 143, Portland, Oregon
  - Local Institution - 179, Germantown, Tennessee
  - Local Institution - 122, Dallas, Texas
- Local Institution - 152, Camperdown, New South Wales, Australia
- Local Institution - 751, Vitebsk, Belarus
- Belgium (2):
  - Local Institution - 600, Ghent
  - Local Institution - 601, Leuven
- Bulgaria (3):
  - Local Institution - 450, Sofia
  - Local Institution - 459, Sofia
  - Local Institution - 451, Sofia
- Local Institution - 264, Lindsay, Ontario, Canada
- Local Institution - 611, Osijek, Croatia
- Czechia (2):
  - Local Institution - 342, Klatovy
  - Local Institution - 337, Prague
- Germany (3):
  - Local Institution - 535, Berlin
  - Local Institution - 525, Berlin
  - Local Institution - 545, Frankfurt
- Local Institution - 643, Athens, Greece
- Hungary (2):
  - Local Institution - 816, Balatonfüred
  - Local Institution - 808, Debrecen
- Local Institution - 505, Rehovot, Israel
- Local Institution - 567, Florence, Tuscany, Italy
- Moldova (2):
  - Local Institution - 658, Chisinau
  - Local Institution - 659, Chisinau
- Local Institution - 425, Kłodzko, Poland
- Romania (2):
  - Local Institution - 677, Bucharest
  - Local Institution - 673, Bucharest
- Local Institution - 910, Bardejov, Slovakia
- South Korea (2):
  - Local Institution - 364, Seongnam-si
  - Local Institution - 354, Wŏnju
- Ukraine (2):
  - Local Institution - 954, Kharkiv
  - Local Institution - 957, Vinnytsia
- United Kingdom (2):
  - Local Institution - 236, London, GREATER LONDON
  - Local Institution - 243, London

REFERENCES:
- [Derived] Yarur A, Irving P, Siegmund B, Dubinsky MC, Ananthakrishnan AN, Regueiro M, Ungaro RC, Ritter T, Nakase H, Liu Z, Mehra D, Osterman MT, Jain A, Rubin DT, Hibi T. Long-Term Ozanimod Therapy in Patients With Moderately Active Ulcerative Colitis After Failure of 5-Aminosalicylic Acid. Inflamm Bowel Dis. 2026 Jan 1;32(1):77-86. doi: 10.1093/ibd/izaf195. PMID 41003640
- [Derived] Sands BE, Rubin DT, Loftus EV Jr, Wolf DC, Panaccione R, Colombel JF, Dignass A, Regueiro M, Vermeire S, Afzali A, Lawlor G, Ahmad HA, Wu H, Osterman MT, Jain A, D'Haens G. Impact of Prior Biologic Exposure on Ozanimod Efficacy and Safety in the Phase 3 True North Clinical Trial. Am J Gastroenterol. 2025 Oct 1;120(10):2339-2349. doi: 10.14309/ajg.0000000000003310. Epub 2025 Jan 8. PMID 39773524
- [Derived] Regueiro M, Siegmund B, Horst S, Moslin R, Charles L, Petersen A, Tatosian D, Wu H, Lawlor G, Fischer M, D'Haens G, Colombel JF. Concomitant Administration of Ozanimod and Serotonergic Antidepressants in Patients With Ulcerative Colitis or Relapsing Multiple Sclerosis. Inflamm Bowel Dis. 2025 Apr 10;31(4):1010-1017. doi: 10.1093/ibd/izae136. PMID 39018016
- [Derived] Sands BE, D'Haens G, Panaccione R, Regueiro M, Ghosh S, Hudesman D, Ahmad HA, Mehra D, Wu H, Jain A, Petersen A, Osterman MT, Afzali A, Danese S. Ozanimod in Patients With Moderate to Severe Ulcerative Colitis Naive to Advanced Therapies. Clin Gastroenterol Hepatol. 2024 Oct;22(10):2084-2095.e4. doi: 10.1016/j.cgh.2024.03.042. Epub 2024 May 8. PMID 38723981
- [Derived] Armuzzi A, Cross RK, Lichtenstein GR, Hou J, Deepak P, Regueiro M, Wolf DC, Akukwe L, Ahmad HA, Jain A, Kozinn M, Wu H, Petersen A, Charles L, Long M. Cardiovascular Safety of Ozanimod in Patients With Ulcerative Colitis: True North and Open-Label Extension Analyses. Clin Gastroenterol Hepatol. 2024 May;22(5):1067-1076.e3. doi: 10.1016/j.cgh.2023.11.018. Epub 2023 Nov 30. PMID 38040274
- [Derived] Sandborn WJ, Feagan BG, Hanauer S, Vermeire S, Ghosh S, Liu WJ, Petersen A, Charles L, Huang V, Usiskin K, Wolf DC, D'Haens G. Long-Term Efficacy and Safety of Ozanimod in Moderately to Severely Active Ulcerative Colitis: Results From the Open-Label Extension of the Randomized, Phase 2 TOUCHSTONE Study. J Crohns Colitis. 2021 Jul 5;15(7):1120-1129. doi: 10.1093/ecco-jcc/jjab012. PMID 33438008
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- RPC01-3101 Placebo-Placebo; RPC01-3101 Ozanimod-Placebo; RPC01-3101 Ozanimod-Ozanimod: Participants who previously participated in RPC01-3101 and met the eligibility criteria received Ozanimod 1 mg daily
- RPC01-202 Ozanimod Open Label: Participants who completed at least 1 year of the open-label period of RPC01-202 for ulcerative colitis and met the eligibility criteria received Ozanimod 1 mg daily
Period: Overall Study
Arm/Group | RPC01-3101 Placebo-Placebo | RPC01-3101 Ozanimod-Placebo | RPC01-3101 Ozanimod-Ozanimod | RPC01-202 Ozanimod Open Label
Started | 184 | 196 | 443 | 54
Completed | 41 | 78 | 135 | 29
Not Completed | 143 | 118 | 308 | 25
Not completed — Non-compliance with protocol/protocol deviation | 5 | 0 | 3 | 0
Not completed — Adverse Event | 16 | 13 | 27 | 4
Not completed — Lack of Efficacy | 50 | 32 | 121 | 0
Not completed — Withdrawal by Subject | 38 | 31 | 96 | 6
Not completed — Pregnancy | 2 | 3 | 2 | 0
Not completed — Switched to commercial drug | 2 | 4 | 4 | 0
Not completed — Other reasons | 23 | 29 | 27 | 15
Not completed — Physician Decision | 6 | 6 | 28 | 0
Not completed — Non-compliance with investigational drug | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RPC01-3101 Placebo-Placebo | RPC01-3101 Ozanimod-Placebo | RPC01-3101 Ozanimod-Ozanimod | RPC01-202 Ozanimod Open Label | Total
Number analyzed (Participants) | 184 | 196 | 443 | 54 | 877
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 171 | 188 | 420 | 54 | 833
  >=65 years | 13 | 8 | 23 | 0 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 91 | 184 | 22 | 357
  Male | 124 | 105 | 259 | 32 | 520
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 11 | 19 | 1 | 37
  Not Hispanic or Latino | 178 | 185 | 424 | 53 | 840
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 13 | 10 | 31 | 3 | 57
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 9 | 11 | 1 | 25
  White | 165 | 174 | 394 | 48 | 781
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 7 | 2 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Treatment-Emergent Adverse Event (TEAEs)
Description: Number of participants experiencing TEAEs, Serious TEAEs, TEAEs leading to discontinuation and TEAEs of special interest. TEAE is defined as any event with an onset date on or after the first dose date, or any ongoing event on the first dose date that worsens in severity on or after the first dose date, and until 90 days following the last dose of treatment with the study drug.
Time Frame: From first dose to 90 days post last dose (Up to approximately 92 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | RPC01-3101 Placebo-Placebo | RPC01-3101 Ozanimod-Placebo | RPC01-3101 Ozanimod-Ozanimod | RPC01-202 Ozanimod Open Label
Number analyzed (Participants) | 184 | 196 | 443 | 54
Participants
  TEAEs | 139 | 160 | 342 | 37
  Serious TEAEs | 24 | 41 | 76 | 8
  TEAE Leading to Discontinuation of Study Drug | 17 | 14 | 33 | 4
  TEAEs of Special Interest | 28 | 32 | 55 | 6

2. Secondary Outcome: Percentage of Participants With Clinical Remission
Description: Clinical Remission is defined as Rectal bleeding subscore=0; stool frequency subscore <=1 (and a decrease of >=1 point from the baseline stool frequency subscore); and endoscopy subscore <=1.
  Rectal bleeding 0 = No blood seen Stool frequency 0 = Normal number of stools for this patient; 1 = 1 to 2 stools more than normal Endoscopy 0 = Normal or inactive disease; 1 = Mild disease (erythema, decreased vascular pattern, does not include friability).
Time Frame: Week 46, 94, 142, 190, 238
Population: All treated participants who are evaluated for clinical remission at the specified visit point
Measure: Number; unit: Percentage of participants
Arm/Group | RPC01-3101 Placebo-Placebo | RPC01-3101 Ozanimod-Placebo | RPC01-3101 Ozanimod-Ozanimod | RPC01-202 Ozanimod Open Label
Number analyzed (Participants) | 113 | 140 | 266 | 0
Percentage of participants
  week 46 | 41.6 | 62.9 | 44.0 |
  week 94: number analyzed (Participants) | 90 | 117 | 202 | 0
  week 94 | 57.8 | 59.0 | 50.5 |
  week 142: number analyzed (Participants) | 69 | 106 | 173 | 0
  week 142 | 59.4 | 60.4 | 50.9 |
  week 190: number analyzed (Participants) | 46 | 77 | 150 | 0
  week 190 | 39.1 | 64.9 | 54.7 |
  week 238: number analyzed (Participants) | 39 | 58 | 112 | 0
  week 238 | 38.5 | 63.8 | 54.5 |

3. Secondary Outcome: Percentage of Participants With Clinical Response
Description: Clinical response is defined as reduction from baseline in the 9-point Mayo score of >=2 points and reduction from baseline in the 9-point Mayo score >=35%, and (reduction from baseline in the rectal bleeding subscore of >=1 point or a rectal bleeding subscore of <=1 point). 9 point Mayo score is defined as the sum of rectal bleeding subscore, stool frequency subscore, and the endoscopy subscore each ranging from (0=normal activity-3=worse activity) for a total score that ranges from 0 to 9 with higher score indicating worsening symptoms.
Time Frame: Week 46, 94, 142, 190, 238
Population: All treated participants who are evaluated for clinical response at the specified visit point
Measure: Number; unit: Percentage of participants
Arm/Group | RPC01-3101 Placebo-Placebo | RPC01-3101 Ozanimod-Placebo | RPC01-3101 Ozanimod-Ozanimod | RPC01-202 Ozanimod Open Label
Number analyzed (Participants) | 110 | 136 | 261 | 0
Percentage of participants
  week 46 | 81.8 | 89.7 | 77.0 |
  week 94: number analyzed (Participants) | 88 | 113 | 199 | 0
  week 94 | 84.1 | 92.9 | 83.9 |
  week 142: number analyzed (Participants) | 67 | 102 | 170 | 0
  week 142 | 89.6 | 90.2 | 87.6 |
  week 190: number analyzed (Participants) | 45 | 76 | 147 | 0
  week 190 | 82.2 | 96.1 | 86.4 |
  week 238: number analyzed (Participants) | 39 | 57 | 111 | 0
  week 238 | 74.4 | 91.2 | 90.1 |

4. Secondary Outcome: Percentage of Participants With Endoscopic Improvement
Description: Endoscopic Improvement is defined as endoscopy subscore of <=1 point. 0 = Normal or inactive disease;
  1. = Mild disease (erythema, decreased vascular pattern, does not include friability)
  2. = Moderate disease (marked erythema, lack of vascular pattern, friability, erosions)
  3. = Severe disease (spontaneous bleeding, ulceration)
Time Frame: Week 46, 94, 142, 190, 238
Population: All treated participants who are evaluated for endoscopic improvement at the specified visit point
Measure: Number; unit: Percentage of participants
Arm/Group | RPC01-3101 Placebo-Placebo | RPC01-3101 Ozanimod-Placebo | RPC01-3101 Ozanimod-Ozanimod | RPC01-202 Ozanimod Open Label
Number analyzed (Participants) | 121 | 150 | 290 | 30
Percentage of participants
  week 46: number analyzed (Participants) | 121 | 150 | 290 | 29
  week 46 | 51.2 | 72.0 | 49.7 | 41.4
  week 94: number analyzed (Participants) | 94 | 127 | 215 | 30
  week 94 | 60.6 | 66.9 | 58.6 | 50.0
  week 142: number analyzed (Participants) | 72 | 112 | 186 | 26
  week 142 | 61.1 | 66.1 | 60.8 | 57.7
  week 190: number analyzed (Participants) | 55 | 87 | 168 | 16
  week 190 | 49.1 | 71.3 | 62.5 | 56.3
  week 238: number analyzed (Participants) | 46 | 75 | 133 | 2
  week 238 | 43.5 | 69.3 | 60.9 | 100

5. Secondary Outcome: Percentage of Participants With Corticosteroid-free Remission
Description: Corticosteroid-free remission is defined as clinical remission while off corticosteroids for ≥12 weeks. Clinical Remission is defined as Rectal bleeding subscore=0; stool frequency subscore <=1 (and a decrease of >=1 point from the baseline stool frequency subscore); and endoscopy subscore <=1.
  Rectal bleeding 0 = No blood seen Stool frequency 0 = Normal number of stools for this patient; 1 = 1 to 2 stools more than normal Endoscopy 0 = Normal or inactive disease; 1 = Mild disease (erythema, decreased vascular pattern, does not include friability).
Time Frame: Week 46, 94, 142, 190, 238
Population: All treated participants who are evaluated for corticosteroid-free remission at the specified visit point
Measure: Number; unit: Percentage of participants
Arm/Group | RPC01-3101 Placebo-Placebo | RPC01-3101 Ozanimod-Placebo | RPC01-3101 Ozanimod-Ozanimod | RPC01-202 Ozanimod Open Label
Number analyzed (Participants) | 113 | 140 | 266 | 0
Percentage of participants
  week 46 | 40.7 | 53.6 | 38.0 |
  week 94: number analyzed (Participants) | 90 | 117 | 202 | 0
  week 94 | 52.2 | 49.6 | 41.6 |
  week 142: number analyzed (Participants) | 69 | 106 | 173 | 0
  week 142 | 55.1 | 55.7 | 45.1 |
  week 190: number analyzed (Participants) | 46 | 77 | 150 | 0
  week 190 | 37.0 | 57.1 | 47.3 |
  week 238: number analyzed (Participants) | 39 | 58 | 112 | 0
  week 238 | 38.5 | 60.3 | 48.2 |

6. Secondary Outcome: Percentage of Participants With Histologic Remission
Description: Histologic remission is defined as Geboes index score < 2.0. The Geboes score is a validated histological grading system for UC that ranges from 0=no disease activity to 5=high disease activity.
Time Frame: Week 46, 94, 142, 190, 238
Population: All treated participants who are evaluated for histologic remission at the specified visit point
Measure: Number; unit: Percentage of participants
Arm/Group | RPC01-3101 Placebo-Placebo | RPC01-3101 Ozanimod-Placebo | RPC01-3101 Ozanimod-Ozanimod | RPC01-202 Ozanimod Open Label
Number analyzed (Participants) | 108 | 141 | 276 | 30
Percentage of participants
  week 46: number analyzed (Participants) | 108 | 141 | 276 | 27
  week 46 | 19.4 | 30.5 | 25.4 | 48.1
  week 94: number analyzed (Participants) | 84 | 121 | 201 | 30
  week 94 | 22.6 | 36.4 | 32.8 | 26.7
  week 142: number analyzed (Participants) | 70 | 106 | 176 | 25
  week 142 | 32.9 | 37.7 | 32.4 | 48.0
  week 190: number analyzed (Participants) | 49 | 83 | 158 | 16
  week 190 | 42.9 | 53.0 | 47.5 | 62.5
  week 238: number analyzed (Participants) | 41 | 70 | 123 | 1
  week 238 | 34.1 | 57.1 | 56.1 | 100

7. Secondary Outcome: Percentage of Participants With Mucosal Healing
Description: Mucosal Healing is defined as Endoscopy subscore of ≤ 1 point (0 = Normal or inactive disease; 1 = Mild disease (erythema, decreased vascular pattern, does not include friability)) and a Geboes index score < 2.0 (The Geboes score is a validated histological grading system for UC that ranges from 0=no disease activity to 5=high disease activity.)
Time Frame: Week 46, 94, 142, 190, 238
Population: All treated participants who are evaluated for mucosal healing at the specified visit point
Measure: Number; unit: Percentage of participants
Arm/Group | RPC01-3101 Placebo-Placebo | RPC01-3101 Ozanimod-Placebo | RPC01-3101 Ozanimod-Ozanimod | RPC01-202 Ozanimod Open Label
Number analyzed (Participants) | 108 | 141 | 276 | 30
Percentage of participants
  week 46: number analyzed (Participants) | 108 | 141 | 275 | 27
  week 46 | 14.8 | 27.0 | 20.4 | 25.9
  week 94: number analyzed (Participants) | 84 | 119 | 200 | 30
  week 94 | 19.0 | 34.5 | 28.0 | 20.0
  week 142: number analyzed (Participants) | 67 | 106 | 175 | 25
  week 142 | 32.8 | 32.1 | 27.4 | 44.0
  week 190: number analyzed (Participants) | 49 | 82 | 157 | 16
  week 190 | 32.7 | 48.8 | 43.9 | 37.5
  week 238: number analyzed (Participants) | 41 | 70 | 123 | 1
  week 238 | 26.8 | 48.6 | 46.3 | 100

8. Secondary Outcome: Change From Baseline in Complete Mayo Score
Description: The Complete Mayo Score is a composite of four assessments, each rated from 0 to 3:
  1. Stool frequency: (0 = Normal number of stools for this patient; 1 = 1 to 2 stools more than normal; 2 = 3 to 4 stools more than normal; 3 = 5 or more stools more than normal)
  2. Rectal bleeding (0 = No blood seen; 1 = Streaks of blood with stool less than half the time; 2 = Obvious blood with stool most of the time; 3 = Blood alone passes)
  3. endoscopy (0 = Normal or inactive disease; 1 = Mild disease; 2 = Moderate disease; 3 = Severe disease)
  4. Physician's Global Assessment (0 = Normal; 1 = Mild disease; 2 = Moderate disease; 3 = Severe disease).
  The total score range is from 0-12, with higher score indicating worse disease activity. Baseline is the last measurement collected on or prior to the date of first dose in the 3102 OLE study.
Time Frame: Baseline, week 46, 94, 142, 190, 238, 286, 334, 382
Population: All treated participants from RPC01-3101 as pre-specified with baseline and post-baseline measurements at the specified time points
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RPC01-3101 Placebo-Placebo | RPC01-3101 Ozanimod-Placebo | RPC01-3101 Ozanimod-Ozanimod
Number analyzed (Participants) | 108 | 132 | 255
Score on a scale
  week 46 | -3.5 (3.06) | -2.9 (3.31) | -1.8 (2.88)
  week 94: number analyzed (Participants) | 84 | 113 | 192
  week 94 | -3.7 (3.30) | -2.7 (3.21) | -2.2 (3.16)
  week 142: number analyzed (Participants) | 67 | 102 | 164
  week 142 | -4.2 (3.42) | -2.7 (3.38) | -2.5 (3.17)
  week 190: number analyzed (Participants) | 45 | 73 | 144
  week 190 | -3.6 (3.37) | -2.3 (3.35) | -2.6 (3.24)
  week 238: number analyzed (Participants) | 38 | 53 | 106
  week 238 | -3.4 (3.30) | -2.6 (3.50) | -2.9 (3.39)
  week 286: number analyzed (Participants) | 15 | 6 | 21
  week 286 | -4.1 (2.99) | -5.2 (3.54) | -3.9 (3.44)
  week 334: number analyzed (Participants) | 2 | 0 | 8
  week 334 | -4.5 (6.36) |  | -4.4 (3.46)
  week 382: number analyzed (Participants) | 0 | 0 | 1
  week 382 |  |  | -4.0 (NA) — insufficient number of participants to calculate standard deviation

9. Secondary Outcome: Change From Baseline in Partial Mayo Score
Description: The Partial Mayo Score is a composite of three assessments, each rated from 0 to 3:
  1. Stool frequency: (0 = Normal number of stools for this patient; 1 = 1 to 2 stools more than normal; 2 = 3 to 4 stools more than normal; 3 = 5 or more stools more than normal)
  2. Rectal bleeding (0 = No blood seen; 1 = Streaks of blood with stool less than half the time; 2 = Obvious blood with stool most of the time; 3 = Blood alone passes)
  3. Physician's Global Assessment (0 = Normal; 1 = Mild disease; 2 = Moderate disease; 3 = Severe disease).
  The total score range is from 0-9, with higher score indicating worse disease activity. Baseline is the last measurement collected on or prior to the date of first dose in the 3102 OLE study.
Time Frame: Baseline, week 46, 94, 142, 190, 238, 286, 334, 382
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RPC01-3101 Placebo-Placebo | RPC01-3101 Ozanimod-Placebo | RPC01-3101 Ozanimod-Ozanimod
Number analyzed (Participants) | 114 | 153 | 281
Score on a scale
  week 46 | -2.8 (2.50) | -2.2 (2.56) | -1.4 (2.20)
  week 94: number analyzed (Participants) | 95 | 133 | 222
  week 94 | -2.9 (2.65) | -2.1 (2.64) | -1.8 (2.35)
  week 142: number analyzed (Participants) | 81 | 119 | 183
  week 142 | -3.1 (2.75) | -2.3 (2.66) | -1.9 (2.31)
  week 190: number analyzed (Participants) | 60 | 91 | 160
  week 190 | -3.0 (2.42) | -2.0 (2.71) | -2.0 (2.39)
  week 238: number analyzed (Participants) | 46 | 66 | 124
  week 238 | -2.8 (2.62) | -2.1 (2.60) | -2.2 (2.61)
  week 286: number analyzed (Participants) | 19 | 7 | 24
  week 286 | -3.5 (2.29) | -3.9 (3.34) | -3.5 (2.70)
  week 334: number analyzed (Participants) | 2 | 0 | 11
  week 334 | -2.5 (6.36) |  | -2.8 (2.60)
  week 382: number analyzed (Participants) | 1 | 0 | 1
  week 382 | -6.0 (NA) — insufficient number of participants to calculate standard deviation |  | -4.0 (NA) — insufficient number of participants to calculate standard deviation

10. Secondary Outcome: Change From Baseline in 9-Point Mayo Score
Description: The 9-point Mayo Score is a composite of three assessments, each rated from 0 to 3:
  1. Stool frequency: (0 = Normal number of stools for this patient; 1 = 1 to 2 stools more than normal; 2 = 3 to 4 stools more than normal; 3 = 5 or more stools more than normal)
  2. Rectal bleeding (0 = No blood seen; 1 = Streaks of blood with stool less than half the time; 2 = Obvious blood with stool most of the time; 3 = Blood alone passes)
  3. Endoscopy (0 = Normal or inactive disease; 1 = Mild disease; 2 = Moderate disease; 3 = Severe disease) The total score range is from 0-9, with higher score indicating worse disease activity. Baseline is the last measurement collected on or prior to the date of first dose in the 3102 OLE study.
Time Frame: Baseline, week 46, 94, 142, 190, 238, 286, 334, 382
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RPC01-3101 Placebo-Placebo | RPC01-3101 Ozanimod-Placebo | RPC01-3101 Ozanimod-Ozanimod
Number analyzed (Participants) | 108 | 132 | 255
Score on a scale
  week 46 | -2.4 (2.31) | -2.1 (2.48) | -1.3 (2.23)
  week 94: number analyzed (Participants) | 84 | 113 | 192
  week 94 | -2.5 (2.48) | -1.8 (2.47) | -1.5 (2.44)
  week 142: number analyzed (Participants) | 67 | 102 | 164
  week 142 | -2.8 (2.66) | -1.8 (2.62) | -1.6 (2.45)
  week 190: number analyzed (Participants) | 45 | 73 | 144
  week 190 | -2.4 (2.61) | -1.5 (2.53) | -1.7 (2.48)
  week 238: number analyzed (Participants) | 38 | 53 | 106
  week 238 | -2.2 (2.52) | -1.6 (2.62) | -2.0 (2.54)
  week 286: number analyzed (Participants) | 15 | 6 | 21
  week 286 | -3.0 (2.33) | -3.5 (2.43) | -2.8 (2.59)
  week 334: number analyzed (Participants) | 2 | 0 | 8
  week 334 | -3.5 (4.95) |  | -3.1 (2.47)
  week 382: number analyzed (Participants) | 0 | 0 | 1
  week 382 |  |  | -3.0 (NA) — insufficient number of participants to calculate standard deviation

11. Secondary Outcome: Percentage of Participants Who Had Previously Received Anti-TNF Therapy With Clinical Remission
Description: as for outcome 2
Time Frame: Week 46, 94, 142, 190, 238
Population: All treated participants who had previously received anti-TNF therapy and who are evaluated for clinical remission at the specified visit point
Measure: Number; unit: Percentage of participants
Arm/Group | RPC01-3101 Placebo-Placebo | RPC01-3101 Ozanimod-Placebo | RPC01-3101 Ozanimod-Ozanimod | RPC01-202 Ozanimod Open Label
Number analyzed (Participants) | 26 | 36 | 266 | 0
Percentage of participants
  week 46: number analyzed (Participants) | 26 | 36 | 86 | 0
  week 46 | 19.2 | 44.4 | 31.4 |
  week 94: number analyzed (Participants) | 15 | 25 | 64 | 0
  week 94 | 46.7 | 52.0 | 43.8 |
  week 142: number analyzed (Participants) | 9 | 21 | 52 | 0
  week 142 | 44.4 | 66.7 | 42.3 |
  week 190: number analyzed (Participants) | 7 | 20 | 43 | 0
  week 190 | 42.9 | 75.0 | 48.8 |
  week 238: number analyzed (Participants) | 7 | 17 | 38 | 0
  week 238 | 28.6 | 58.8 | 47.4 |

12. Secondary Outcome: Percentage of Participants Who Had Previously Received Anti-TNF Therapy With Clinical Response
Description: as for outcome 3
Time Frame: Week 46, 94, 142, 190, 238
Population: All treated participants who had Previously Received anti-TNF Therapy and who are evaluated for clinical response at the specified visit point
Measure: Number; unit: Percentage of participants
Arm/Group | RPC01-3101 Placebo-Placebo | RPC01-3101 Ozanimod-Placebo | RPC01-3101 Ozanimod-Ozanimod | RPC01-202 Ozanimod Open Label
Number analyzed (Participants) | 110 | 136 | 261 | 0
Percentage of participants
  week 46: number analyzed (Participants) | 25 | 35 | 85 | 0
  week 46 | 64.0 | 71.4 | 74.1 |
  week 94: number analyzed (Participants) | 14 | 24 | 63 | 0
  week 94 | 64.3 | 95.8 | 84.1 |
  week 142: number analyzed (Participants) | 8 | 20 | 51 | 0
  week 142 | 75.0 | 90.0 | 84.3 |
  week 190: number analyzed (Participants) | 7 | 20 | 42 | 0
  week 190 | 85.7 | 95.0 | 88.1 |
  week 238: number analyzed (Participants) | 7 | 17 | 37 | 0
  week 238 | 71.4 | 76.5 | 86.5 |

13. Secondary Outcome: Percentage of Participants Who Had Previously Received Anti-TNF Therapy With Endoscopic Improvement
Description: Endoscopic Improvement is defined as endoscopy subscore of <=1 point. 0 = Normal or inactive disease;
  1 = Mild disease (erythema, decreased vascular pattern, does not include friability)
Time Frame: Week 46, 94, 142, 190, 238
Population: All treated participants who had Previously Received anti-TNF Therapy and who are evaluated for endoscopic improvement at the specified visit point
Measure: Number; unit: Percentage of participants
Arm/Group | RPC01-3101 Placebo-Placebo | RPC01-3101 Ozanimod-Placebo | RPC01-3101 Ozanimod-Ozanimod | RPC01-202 Ozanimod Open Label
Number analyzed (Participants) | 121 | 150 | 290 | 30
Percentage of participants
  week 46: number analyzed (Participants) | 28 | 38 | 96 | 2
  week 46 | 28.6 | 55.3 | 37.5 | 50.0
  week 94: number analyzed (Participants) | 16 | 27 | 66 | 3
  week 94 | 50.0 | 66.7 | 56.1 | 33.3
  week 142: number analyzed (Participants) | 10 | 21 | 58 | 4
  week 142 | 40.0 | 76.2 | 56.9 | 75.0
  week 190: number analyzed (Participants) | 10 | 22 | 49 | 1
  week 190 | 60.0 | 81.8 | 57.1 | 100
  week 238: number analyzed (Participants) | 7 | 21 | 43 | 0
  week 238 | 42.9 | 61.9 | 60.5 |

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from first dose until study completion (up to approximately 108 months). SAEs and Other AEs were assessed from first dose through 90 days following last dose of study treatment (Up to approximately 92 months)
Arm/Group | RPC01-3101 Placebo-Placebo | RPC01-3101 Ozanimod-Placebo | RPC01-3101 Ozanimod-Ozanimod | RPC01-202 Ozanimod Open Label
All-Cause Mortality (participants affected / at risk) | 0/184 | 0/196 | 3/443 | 0/54
Serious Adverse Events (participants affected / at risk) | 24/184 | 41/196 | 76/443 | 8/54
Other Adverse Events (participants affected / at risk) | 98/184 | 121/196 | 245/443 | 24/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RPC01-3101 Placebo-Placebo (N=184) | RPC01-3101 Ozanimod-Placebo (N=196) | RPC01-3101 Ozanimod-Ozanimod (N=443) | RPC01-202 Ozanimod Open Label (N=54)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 1 | 0
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Congenital anomaly in offspring (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0
Ulcerative keratitis (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 3 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 8 | 8 | 13 | 2
Colon dysplasia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders and administration site conditions) | 0 | 2 | 0 | 0
Hyperthermia (General disorders and administration site conditions) | 0 | 0 | 1 | 0
Pyrexia (General disorders and administration site conditions) | 0 | 0 | 1 | 0
Sudden death (General disorders and administration site conditions) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 2 | 0
Biliary sepsis (Infections and infestations) | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 3 | 4 | 3 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 4 | 5 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 0
Keratouveitis (Infections and infestations) | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0
West Nile viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Colorectal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Follicular lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Rectal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Hemihypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Hemiplegia (Nervous system disorders) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 2 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Parkinsonism (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Large intestine anastomosis (Surgical and medical procedures) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RPC01-3101 Placebo-Placebo (N=184) | RPC01-3101 Ozanimod-Placebo (N=196) | RPC01-3101 Ozanimod-Ozanimod (N=443) | RPC01-202 Ozanimod Open Label (N=54)
Anaemia (Blood and lymphatic system disorders) | 17 | 8 | 32 | 3
Leukopenia (Blood and lymphatic system disorders) | 8 | 8 | 16 | 4
Lymphopenia (Blood and lymphatic system disorders) | 31 | 34 | 72 | 9
COVID-19 (Infections and infestations) | 15 | 33 | 50 | 14
Nasopharyngitis (Infections and infestations) | 9 | 16 | 34 | 3
Upper respiratory tract infection (Infections and infestations) | 8 | 15 | 20 | 0
Alanine aminotransferase increased (Investigations) | 17 | 17 | 30 | 2
Gamma-glutamyltransferase increased (Investigations) | 11 | 20 | 20 | 3
Lymphocyte count decreased (Investigations) | 19 | 25 | 48 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 11 | 30 | 1
Headache (Nervous system disorders) | 8 | 9 | 25 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 12 | 17 | 2
Hypertension (Vascular disorders) | 6 | 18 | 25 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT02531126/Prot_SAP_000.pdf